CLINICAL TRIAL: NCT02915757
Title: Naturalistic Clinical Studies in Several Centres of Electrodermal Hyporeactivity in Adult Patients With Primary Depression
Brief Title: Electrodermal Hyporeactivity And Depression
Acronym: EUDOR-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University of Molise (Other); EMOTRA-AB, Göteborgsvagen 74, 433 63 Sävedalen, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UF 9464; 2014-A01310-47 (Other: Agence Nationale de sécurité des Médicaments)
Record Dates: First submitted 2016-07-20; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-07

CONDITIONS: Depression Diagnosis
Keywords: Depression; EDOR test; Electrodermal hyporeactivity
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Depressive patients (Experimental): EDOR test on depressed patients with or without personal history of suicidal behavior
  Interventions: Device: EDOR test

INTERVENTIONS:
Device: EDOR test — The ElectroDermal Orienting Reactivity (EDOR) specifically is optimized for the detection of electrodermal hyporeactivity.
  The EDOR investigation last about 30 min. The EDOR Test Data is sent immediately after each EDOR Test for each Test Person to a Company named EMOTRA for blind analyses. The EDOR Test Report may change the basis for the assessment and a new risk assessment may be needed to be done.
  Blood sample and clinical assessment

SUMMARY:
Suicide, suicide attempts and depression are major social problems. The present research program focuses on the relationship between electrodermal hyporeactivity, as measured by the ElectroDermal Orienting Reactivity (EDOR) Test, and suicide and suicide attempts with death intent in patients with a primary diagnosis of depression. Electrodermal hyporeactivity has in several publications from different laboratories repeatedly been shown to have a high sensitivity (up to 97%) and high raw specificity (up to 98%) for suicide. Such levels are unique in psychiatry. The relationship between suicidal propensity and hyporeactivity can be considered as strongly significant. Almost all evidence in the topic up today has been established in research settings with specific exclusion criteria for some secondary psychiatric and some somatic illnesses. However, it is important to study the relationship between electrodermal hyporeactivity and suicide in relatively unselected patients regarding secondary psychiatric diagnoses and somatic diagnoses in a natural clinical ward situation and milieu. A previous naturalistic study proved that a test of electrodermal hyporeactivity fits very well into the daily clinical work.

DETAILED DESCRIPTION:
This EUDOR-A study is a naturalistic, european and multicentric study. In France, patient's recruitment will be only conducted by investigators within the Department of Psychiatric Emergencies and Post Acute Care, University Hospital of Montpellier.

Over one year, 233 patients suffering from a major depressive episode with (n=70) and without any history of suicide attempt (n=163) will be recruited.

The maximum period of participation for a given patient will be 12 months with 2 phone assessments at 6 month and 12 month.

Inclusion visit: clinical and biological assessment and Edor test. Second and third visits at 6 and 12 month: Follow up visits in the department or interview by telephone in order to assess suicidal ideations or suicide attempts since the inclusion.

ELIGIBILITY:
Inclusion criteria:

All subjects men and women will necessarily meet the following inclusion criteria:

* In- and outpatients, with a diagnosis of primary depression according to the International classification of Disease (ICD-10) should be included as a routine. That is, patients in a primary unipolar major episode or dysthymia or primary depression with a personality disorder or an anxiety disorder as secondary diagnoses and primary bipolar disorder in a non-hypomanic and non-manic phase are expected to be included.
* Age : 18 years or older
* written informed consent
* must belong to social safety system
* To be able to understand instructions for the EDOR Test, the aim and the methodology of the study.

Exclusion criteria:

* diagnosed or suspected dementia
* Acute known or suspected alcohol or other substance abuse. The condition of past substance abuse (i.e. alcohol abuse or dependance, drug abuse or dependance ) should be noted in the comment field of the EDOR Test routine and patient must have been abstinent for at least one year.
* Serious problems of hearing, the patient should not participate.
* Refusal of participation
* Subject deprived of liberty (by judicial or administrative decision)
* Subject protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Specificity and sensibility of the electrodermal hyporeactivity | At 6 and 12 month
  Correlation between the Edor Test results and suicidal behavior

SECONDARY OUTCOMES:
The sensibility of the electrodermal hyporeactivity compared with the occurrence of the violent suicidal attempt measured by Columbia-Suicide Severity Rating Scale (C-SSRS) | At 6 month
  Comparison of test result between patients with history of violent suicidal attempt and patients with history of non violent suicidal
The sensibility of the electrodermal hyporeactivity compared with the occurrence of the violent suicidal attempt measured by Columbia-Suicide Severity Rating Scale (C-SSRS) | At 6 and 12 month
  Comparison of test result between patients with history of violent suicidal attempt and patients with history of non violent suicidal
Electrodermal activity in depressive and suicidal patients with or without insomnia. | At 6 and 12 month
  Comparison of test result between patients with insomnia and patient without insomnia. Insomnia will be evaluated with the "Insomnia severity index" (ISI).
Genetic vulnerability to suicidal behavior by polymorphism analysis in blood sample | At the inclusion
  To study the polymorphisms by blood sample analysis of the promotor of Spermidine/Spermine Acetyltransferase 1 (SAT1), Phenylethanolamine N-Methyltransferase (PNMT) and Noradrenalin Transporter (NAT). between depressed patients with suicidal behavior and depressed patients without suicidal behavior.
The sensibility of the electrodermal hyporeactivity compared with the occurrence of the violent suicidal attempt measured by Risk Rescue Rating Scale (RRRS) | At 6 and 12 month
  Comparison of test result between patients with history of violent suicidal attempt and patients with history of non violent suicidal
The sensibility of the electrodermal hyporeactivity compared with the occurrence of the violent suicidal attempt measured by Beck Scale for Suicidal Intent (SIS). | At 6 and 12 month
  Comparison of test result between patients with history of violent suicidal attempt and patients with history of non violent suicidal

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No